CLINICAL TRIAL: NCT04656106
Title: A Retrospective Multi-centre Non-interventional Study Investigating the Clinical Parameters Associated With the Use of Ryzodeg® (Insulin Degludec/Insulin Aspart) in a Real-world Adult Population With Type 2 Diabetes in South Korea
Brief Title: A Study Investigating the Clinical Parameters Associated With the Use of Ryzodeg® (Insulin Degludec/Insulin Aspart) in a Real-world Adult Population With Type 2 Diabetes in South Korea
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4653; U1111-1257-2534 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ryzodeg: Patients treated with any basal-insulin or premix-insulin for at least 26 weeks prior to switching to Ryzodeg® and treated for at least 26 weeks after switching to Ryzodeg®.
  Interventions: Drug: Ryzodeg®

INTERVENTIONS:
Drug: Ryzodeg® — All patients have been treated at the discretion of the treating physician in accordance with the Ryzodeg® label in South Korea. Hence independently of this study, the treating physician has determined the starting dose of Ryzodeg® as well as any dose adjustments thereafter.

SUMMARY:
This is a non-interventional (observational), retrospective medical record review study collecting data reported in medical records of patients with T2D (Type 2 Diabetes ) who were treated with any basal-insulin or premix-insulin (plus/minus OAD (Oral Antidiabetic Drug)) for at least 26 weeks prior to switching to Ryzodeg® and treated for at least 26 weeks after switching to Ryzodeg® (plus/minus OAD).

All patients have been treated at the discretion of the treating physician in accordance with the Ryzodeg® label in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 19 years at the time of Ryzodeg® initiation
* Type 2 diabetes mellitus patients
* Treated with any basal-insulin (plus/minus OAD (Oral Antidiabetic Drug)) or premix-insulin (plus/minus OAD) for at least 26 weeks prior to switching to Ryzodeg®
* Treated with Ryzodeg® (plus/minus OAD) for at least 26 weeks after switch from any basal insulin (plus/minus OAD) or premix insulin (plus/minus OAD)
* At least more than once documented medical visit for 26weeks (plus/minus 6 weeks) after Ryzodeg® initiation
* Minimum available data : age, type of diabetes at the time of Ryzodeg® initiation, HbA1c [Three values: most recent value within 26 weeks (plus/minus 6 weeks) prior to Ryzodeg® initiation, a value of Ryzodeg® initiation date (plus/minus 6 week), and a value in the first 26 weeks (plus/minus 6 weeks) after Ryzodeg® initiation]
* The decision to treat with Ryzodeg® was taken by treating physician independently from decision to include patient in study.

Exclusion Criteria:

* Patients treated with any diabetic investigational drug within 26 weeks before or after the initiation of Ryzodeg®
* Patients switching to Ryzodeg® below 26 weeks prior to the data collection date
* Patients not treated with any basal-insulin or premix-insulin at least 26 weeks prior to receiving Ryzodeg®
* Patients treated by continuous subcutaneous insulin infusion prior to receiving Ryzodeg®
* Pregnancy patient
* Patients not treated with the local licensed Ryzodeg®

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with any basal-insulin or premix-insulin for at least 26 weeks prior to switching to Ryzodeg® and treated for at least 26 weeks after switching to Ryzodeg®.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (Glycosylated Hemoglobin) | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  Percentage point

SECONDARY OUTCOMES:
Patients with HbA1c less than 7.0 percentage (Yes or No) | At baseline (week 0)
  Percentage of patients
Patients with HbA1c less than 7.0 percentage (Yes or No) | End of study (week 26)
  Percentage of patients
Patients with HbA1c less than 7 percentage without any hypoglycaemic events during the previous 26 weeks (Yes or No) | At baseline (week 0)
  Percentage of patients
Patients with HbA1c less than 7 percentage without any hypoglycaemic events during the previous 26 weeks (Yes or No) | End of study (week 26)
  Percentage of patients
Difference in the number of overall hypoglycaemia events within 26 weeks before and after the switch to Ryzodeg® | Period 1(week-26 to week 0), Period 2(week 0 to week 26)
  Number of events
Difference in the number of severe hypoglycaemia events within 26 weeks before and after the switch to Ryzodeg® | Period 1(week-26 to week 0), Period 2(week 0 to week 26)
  Number of events
Change in FPG (Fasting Plasma Glucose) | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  mmol/L
Change in daily total insulin dose | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  Unit/day
Change in daily basal insulin dose | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  Unit/day
Change in daily prandial insulin dose | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  Unit/day
Change in body weight | Period 1 (week -26 to week 0), Period 2 (week 0 to week 26)
  Kg

CONTACTS AND LOCATIONS:
Overall Officials: Clinical transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (4):
- South Korea (4):
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Kang S, Ahn YB, Oh TK, Lee WY, Chun SW, Bae B, Dahaoui A, Jeong JS, Jung S, Jang HC. Efficacy and Safety of IDegAsp in a Real-World Korean Population with Type 2 Diabetes Mellitus. Diabetes Metab J. 2024 Sep;48(5):929-936. doi: 10.4093/dmj.2023.0297. Epub 2024 Feb 27. PMID 38410023